CLINICAL TRIAL: NCT07207824
Title: A Phase III Randomized Controlled Trial of Disitamab Vedotin (DV) Combined With Bacillus Calmette-Guérin (BCG) in BCG-Naïve Patients With HER2-Expressing, High-Risk Non-Muscle-Invasive Bladder Cancer
Brief Title: DV+BCG in HER2-Expressing, BCG-Naïve High-Risk NMIBC
Acronym: HERO
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Collaborators: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other); Fujian Cancer Hospital (Other Government); Tenth People's Hospital of Tongji Univeristy (Unknown); Ningbo Medical Center Li Huili Hospital (Unknown)
Responsible Party: Principal Investigator, Ding-Wei Ye, Director of Urology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RCVDUCIIR020-2
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Bladder (Urothelial, Transitional Cell) Cancer; NMIBC
Keywords: NMIBC; disitamab vedotin; HER2; BCG
MeSH Terms: conditions — Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Maintenance

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DV + BCG (Experimental): Disitamab Vedotin + BCG induction and maintenance
  Interventions: Drug: DV + BCG induction and maintenance
- BCG (Active Comparator): BCG induction and maintenance
  Interventions: Drug: Active Comparator: BCG induction and maintenance

INTERVENTIONS:
Drug: Active Comparator: BCG induction and maintenance — Drug: Bacillus Calmette-Guerin Immunotherapy treatment approved by NMPA for patients with high-risk non-muscle invasive bladder cancer
  Other Names:
  BCG
  Arms: BCG
Drug: DV + BCG induction and maintenance — Drug: Disitamab vedotin(RC48) •An antibody-drug conjugates (ADCs) targeting HER2, has been approved in China for chemotherapy-refractory advanced UC with HER2-expression.
  Other Names:
  • RC48, DV
  Drug: Bacillus Calmette-Guerin Immunotherapy treatment approved by NMPA for patients with high-risk non-muscle invasive bladder cancer
  Other Names:
  BCG
  Arms: DV + BCG

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine (Disitamab Vedotin) in people with non-muscle invasive bladder cancer. This study is seeking participants whose bladder cancer is still in early stages, has not spread outside of the bladder, has been removed with surgery, and is high risk. Each participant was assigned to one of two study treatment groups: One group is given Disitamab Vedotin and BCG.The second group is given BCG only and will not receive Disitamab Vedotin.

DETAILED DESCRIPTION:
HERO: A Phase III Randomized Controlled Trial of Disitamab Vedotin (DV) Combined with Bacillus Calmette-Guérin (BCG) in BCG-Naïve Patients with HER2-Expressing, High-Risk Non-Muscle-Invasive Bladder Cancer

This Phase 3, open-label, randomized, controlled clinical trial will enroll approximately 182 patients, who will be assigned in a 1:1 ratio to one of two treatment groups:

Group A: Disitamab Vedotin plus BCG (induction and maintenance therapy)

Group B: BCG alone (induction and maintenance therapy)

The study is designed to demonstrate the superiority of Disitamab Vedotin combined with BCG (during both induction and maintenance phases) over BCG alone in prolonging event-free survival (EFS) among BCG-naïve participants with high-risk, HER2-expressing non-muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18 years.
2. Histologically confirmed high-risk, non-muscle-invasive urothelial carcinoma of the bladder (UCC) (with >50% urothelial carcinoma as the predominant histological component), defined by the presence of any of the following: a. T1 tumor; b. High-grade Ta tumor; c. Carcinoma in situ (CIS).
3. Complete resection of all Ta/T1 papillary lesions (including patients with concomitant CIS). The most recent Transurethral Resection of Bladder Tumor (TURBT) must have been performed within 12 weeks prior to randomization. A second TURBT was required if indicated per current local applicable guidelines.
4. HER2 expression (IHC 1+/2+/3+) as confirmed by immunohistochemistry (IHC) testing at the local institution's pathology department.
5. Unwillingness or ineligibility to undergo radical cystectomy.
6. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2.
7. Signed informed consent form (ICF).

Exclusion Criteria

1. Histologically confirmed evidence of muscle-invasive (T2 or higher), locally advanced, or metastatic urothelial carcinoma, or the presence of concurrent extravesical non-muscle-invasive urothelial carcinoma.
2. Histopathological findings of pure small cell carcinoma, pure adenocarcinoma, pure squamous cell carcinoma, or pure squamous CIS of the bladder.
3. History of upper tract urothelial carcinoma (except for cases with no recurrence within 2 years following radical treatment for UTUC).
4. Prior therapy with any other type of HER2-targeted inhibitor.
5. Major surgery within 2 weeks prior to randomization.
6. Any other condition that, in the investigator's judgment, would make the patient unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2030-06-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Event free survival | 55 months after first participant randomized
  Event free survival is defined as the time from randomization to date of EFS event.

SECONDARY OUTCOMES:
Overall Survival | Randomization up to 60 months from last participant randomized
  Overall survival is defined as the time from the date of randomization to the date of death due to any cause.
Complete response rate at 6m/12m in participants with CIS at randomization | Randomization up to 12 months from last participant randomized
  Complete response (CR) rate defined as the proportion of participants in the analysis population with CR.
Disease-specific survival | Randomization up to 60 months from last participant randomized
  Disease specific survival (DSS) is defined as the time from randomization to death resulting from bladder cancer.
Health-related quality of life as measured by EORTC QLQ-C30 | Randomization up to 60 months from last participant randomized
  Health-related quality of life as measured by EORTC QLQ-C30
Health-related quality of life as measured by EORTC QLQ-NMIBC24 | Randomization up to 60 months from last participant randomized
  EORTC-QLQ-NMIBC24 has 24 items which can be grouped into 6 subscales: urinary symptoms (7 items), malaise (2 items), future worries (4 items), bloating/flatulence (2 items), sexual functioning (2 items), and male sexual issues (2 items). The NMIBC24 also assesses intravesical treatment, female sexual issues, sexual intimacy, risk of contaminating a partner, and sexual enjoyment (1 item each).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data is protected.